CLINICAL TRIAL: NCT03386396
Title: Morning Nutrition and Cognitive Function in Preadolescents
Brief Title: Brain Fuel - Morning Nutrition and Cognitive Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 206464
Record Dates: First submitted 2017-12-06; First posted 2017-12-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obese; Healthy
MeSH Terms: conditions — Obesity | interventions — Diet, High-Protein Low-Carbohydrate

STUDY DESIGN:
Intervention Model Description: One group will be given a high protein/low carbohydrate shake and one group will be given a high carbohydrate/low protein shake
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High protein/low carbohydrate (Experimental): A breakfast shake will be made with high protein/low carbohydrate mixture.
  Interventions: Dietary Supplement: High protein/low carbohydrate
- High carbohydrate/low protein (Experimental): A breakfast shake will be made with high carbohydrate/low protein mixture.
  Interventions: Dietary Supplement: High carbohydrate/low protein

INTERVENTIONS:
Dietary Supplement: High protein/low carbohydrate — A high protein/low carbohydrate shake will be given to the child.
  Arms: High protein/low carbohydrate
Dietary Supplement: High carbohydrate/low protein — A high carbohydrate/low protein shake will be given to the child
  Arms: High carbohydrate/low protein

SUMMARY:
This study will help us learn more about how what a child eats can affect how their brain works.

DETAILED DESCRIPTION:
Following a high protein/low carbohydrate meal brain activation and performance measurements will differ from those following a high carbohydrate/low protein meal and executive functioning will be affected.

ELIGIBILITY:
Inclusion Criteria:

* 9-10 yr, 3rd to 5th grade
* Obese
* Right hand dominance
* Report eating breakfast at least 4 days/week
* Able to hear at least 20dB stimulus
* Visual acuity must be at least 20/40
* Biological mother available to attend visit

Exclusion Criteria:

* Full scale IQ <80
* Children taking medications or having chronic illness/disorders

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Psychological assessments | 9-10 years
  Standardized testing

SECONDARY OUTCOMES:
Neurocognitive measures | 9-10 years
  Brain Lab recordings and fMRI readings

CONTACTS AND LOCATIONS:
Overall Officials: Linda Larson-Prior, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States